CLINICAL TRIAL: NCT02893904
Title: Electroencephalographic Profiles During General Anesthesia : a Comparative Study Between Sevoflurane and Propofol.
Brief Title: EEG Profiles During General Anesthesia : a Comparative Study Between Sevoflurane and Propofol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Armand Trousseau (Other)
Collaborators: Club d'Anesthésie-Réanimation Pédiatrique Armand Trousseau (Other)
Responsible Party: Principal Investigator, Pr Isabelle CONSTANT, Pr Isabelle CONSTANT, Hôpital Armand Trousseau
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: BIS and EEG
Record Dates: First submitted 2016-01-21; First posted 2016-09-09 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Anesthesia
Keywords: Propofol; Sevoflurane; Bispectral Index; Children; Electroencephalographic signs

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Experimental): General anesthesia by TCI Propofol and Remifentanil guided by BIS EEG monitoring intervention
  Interventions: Device: EEG monitoring; Device: Target Controlled Infusion
- Sevoflurane (Experimental): General anesthesia by Sevoflurane and Remifentanil guided by BIS EEG monitoring intervention
  Interventions: Device: EEG monitoring; Device: Target Controlled Infusion

INTERVENTIONS:
Device: EEG monitoring — Steady state concentrations periods of Propofol for EEG data analyzes. Remifentanil was administrated at constant rate in all patients.
Device: Target Controlled Infusion — Steady state effect site concentrations of remifentanil administrated to all patients.
  Other Names: TCI

SUMMARY:
A cerebral pharmacodynamic feedback may help the anesthesiologist to adjust anesthetics administration. The BIS, which provides a single number resulting from an algorithm calculated from cortical EEG parameters, may play this role.Moreover, halogenated agents and propofol may have different EEG effects, which might interfere on measured BIS values.

The aim of this prospective randomized study was to compare, in steady state conditions, the EEG profiles in children anesthetized with sevoflurane (S) or propofol (P) : for both anesthetics, the BIS-concentration relationship and raw EEG were analysed at different levels of general anesthesia.

DETAILED DESCRIPTION:
Children will be prospectively included and randomly assigned in two groups : Propofol (P) Group or Sevoflurane (S) Group.

Steady state periods will be performed at a fixed randomized concentration between 2, 3, 4, 5 and 6 mcg/ml of stable Ct P concentration in the P group and between 1,2,3,4,5 % of FeS in the S group.

At the end of each steady-state period the BIS value was noted and the relationship between BIS and anesthetic concentrations will be studied using non linear regression. For all steady state periods, EEG traces will be reviewed to determine the presence of epileptiform signs (ES) and spectral EEG signal analysis with fast Fourier transformation (FFT) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* from five to eighteen year of age, ASA 1 or 2, scheduled for middle ear surgery

Exclusion Criteria:

* obesity (body mass index > percentile 97); history of cardiac, pulmonary, or renal disease; known neurological or neuromuscular disorders; preoperative administration of medications known to interfere with the central nervous system

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 73 (Actual)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Bispectral profiles | The average value of BIS is calculated on the last minute of each ten minutes steady state period .
  For each patient, before surgery and according to the constraints of operating schedule, one or two 10 min steady state periods were performed at a fixed FeS randomized between 1, 2, 3, 4 and 5 % of Sevoflurane in the Sevoflurane group or at a fixed Ct P randomized between 2, 3, 4, 5 and 6 mcg/ml in the propofol group.

SECONDARY OUTCOMES:
Incidence of epileptiform EEG signs | Last minute of each ten minutes steady state period
Spectral analysis of EEG signal | Last minute of each ten minutes steady state period

CONTACTS AND LOCATIONS:
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No